CLINICAL TRIAL: NCT03735511
Title: A Real World Study of Apatinib in Treatment of Patients With Gastric Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: APA-GC-2018-HNZL
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was designed to evaluate the efficacy and safety of apatinib in the treatment of patients with gastric carcinoma.

DETAILED DESCRIPTION:
The study is a real-world non-interventional retrospective study and will collect the original medical records of patients with gastric carcinoma treated with apatinib from 2015 to 2018 in Henan Cancer Hospital. Clinical data such as patient demographic, history of treatments, tumor biological characteristics and adverse events will be analyzed to evaluate the efficacy and safety of apatinib and explore the risk factors of prognosis in patients with gastric carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed gastric or residual gastric or gastroesophageal junction carcinoma;
2. Patients received apatinib treatment at least once.

Exclusion Criteria:

1. No specific exclusion criteria in this real world study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients who were pathologically or cytologically diagnosed gastric carcinoma and treated by apatinib.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2015-2018
  Overall Survival

SECONDARY OUTCOMES:
Objective Response Rate | 2015-2018
  Objective Response Rate
Disease Control Rate | 2015-2018
  Disease Control Rate
Progression-Free Survival | 2015-2018
  Progression-Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No